CLINICAL TRIAL: NCT06513039
Title: Evaluation of Erythropoietin on Alveolar Ridge Preservation: (A Randomized Controlled Clinical Trial With Histomorphometric Assessment)
Brief Title: Evaluation of Erythropoietin on Alveolar Ridge Preservation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, shehad wael, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1111 phd
Record Dates: First submitted 2024-07-14; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Three group randomized clinical trial study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group (Experimental): Patient will have extraction of teeth and placement of Erythropoietin carried on chitosan carrier for six months
  Interventions: Drug: Erythropoietin carried on chitosan carrier
- control (No Intervention): Patient will have extraction of teeth only and followup
- positive control (Active Comparator): Patient will have extraction of teeth and placement of chitosan carrier only for six months
  Interventions: Other: chitosan carrier

INTERVENTIONS:
Drug: Erythropoietin carried on chitosan carrier — Patient will have extraction of teeth and placement of Erythropoietin carried on chitosan carrier for six months to enhance bone healing
  Arms: study group
Other: chitosan carrier — inert scaffold agent
  Arms: positive control

SUMMARY:
regenerative materials would help in decreasing post-extraction resorption in sites indicated for placement of a conventional bridge or prosthetically driven implant. Erythropoietin (EPO) is a growth factor that promotes angiogenesis and bone regeneration by stimulating osteoblastic differentiation and by inhibiting osteoclastic resorption. Post-extraction alveolar ridge resorption creates morphological and volumetric changes. These changes can be considered of clinical value that may threaten the placement of a conventional bridge or an implant-supported crown. Atwood et al. [1] in a cephalometric study categorized factors influencing the rate of alveolar ridge resorption into 4 types: anatomic, metabolic, functional, and prosthetic. As stated by Tan et al. [2] in a systematic review of alveolar hard and soft tissue dimensional changes in humans post-extraction, they found that alveolar ridge resorption occurs to a greater extent in a horizontal direction than vertical. Therefore, alveolar ridge preservation (ARP) procedures were introduced in an attempt to prevent hard and soft tissue dimensional changes following extraction.

DETAILED DESCRIPTION:
II. Aim of the study:

To assess the efficiency of Erythropoietin in alveolar ridge preservation.

1. Objectives:

Primary objective:

Dimensional changes of the ridge clinically and radiographically.

Secondary objective:

1. Postoperative pain.
2. Postoperative wound healing.
3. Histomorphometric analysis of the bone regeneration patterns of the extraction sockets.

III. Materials and Methods

1. Study design and patient selection:

   It is a randomized controlled clinical trial. Patients will be selected from the outpatient clinic of the Department of Oral Medicine and Periodontology-Ain Shams University and the British University of Egypt. All patients will sign an informed consent about the details of the surgery according to the Ethical Committee Ain Shams University.
2. Sample size:

   The sample size was estimated based on assuming confidence level= 95% and study power= 80%. Pandya et al. [29] reported that the Collagen percentage was 2.1%±0.6% in EPO treated sockets while it was 1%±0.6% in non-treated sockets, the average Standard deviation was 0.6%n. The minimum sample size was calculated to be 5 extraction sockets per group. This was increased to 7 sockets to make up for lost to follow-up cases. The total sample size = number of groups × number per group= 3×7= 21 sockets. The sample size was collected by G power 3.0.10.
3. Eligibility criteria:

Inclusion criteria:

1. Age range (18-40).
2. Hopeless teeth indicated for extraction such as root fractures, caries, internal root resorption, external root resorption, endodontic failures.
3. Systemically free patients using Cornell Medical Index-Health Questionnaire [36].
4. Patients diagnosed with intact surrounding alveolar bone (socket type I) [37].
5. Maxillary anterior teeth and/or premolars indicated for extraction.
6. Enough zone of keratinized tissue (≥2 mm).

Exclusion criteria:

1. Smokers
2. Occlusal trauma at the site of the graft
3. Pregnancy and lactation
4. Bad compliance with the plaque control instructions following initial therapy.

4. Interventions:

Pre-surgical phase:

Patients will be initially examined. All patients will receive oral hygiene instructions using roll technique with a soft-bristled toothbrush and interdental floss, and phase I therapy using an ultrasonic device if necessary. At baseline, intraoral periapical radiographs, clinical periodontal measurements including plaque Index [38] , bleeding on probing (BOP) [38], probing depth (PD) [38], and clinical attachment level (CAL) [38] will be recorded at teeth adjacent to the extraction socket area using a UNC periodontal probe [38].

Impressions will be taken using Alginate impression material before the extraction day. Diagnostic casts will be made for the fabrication of a customized stent to standardize the measurements of marginal crestal bone levels at baseline and 4 months post-extraction [39].

Surgical preparation of Extraction socket:

1. After anesthetizing the surgical field with local anesthesia (4% Articaine , 1: 100 000 epinephrine), An atraumatic extraction procedure will be performed by cutting the periodontal ligaments gently to preserve the buccal plate of bone using periotome and forceps.
2. The socket will be irrigated with saline and curetted from any granulation tissue following extraction then the buccal and lingual plate of bone will be checked for absence of any fenestration or dehiscence using UNC periodontal probe.
3. Computer-generated randomization will be used to randomly divide the sockets into three groups. Group I: Extraction sockets filled with CS/ β-GP/gelatin hydrogels loaded EPO until the crestal level.

   Group II: extraction sockets filled with CS/ β-GP/gelatin hydrogels alone until the crestal level.

   Group III: Natural healing socket (control group).
4. In the three groups, the flaps will be sutured with criss-cross horizontal mattress technique with polypropylene 5-0 .

Implant placement Surgery

Patients will return for a follow-up examination at 4 months and implant placement.

1. After anesthetizing the surgical field with local anesthesia (4% Articaine, 1: 100 000 epinephrine), a papillary sparing will be incised using Bard-Parker scalpel carrying blade number 15C; a crestal flap will be elevated by Molt number 5 mucoperiosteal elevator.
2. The first drill will be a trephine bur to collect a core bone biopsy; the collected bone will be preserved in a diluted formaldehyde solution to fix the sample to perform the histomorphometry.
3. Sequential twist drills will be used until the final drill following the implant manufacturer instructions.
4. In the three groups, the flaps will be sutured with criss-cross horizontal mattress technique suture type using 5-0 polypropylene sutures.

Postoperative care instruction and medication of both surgeries:

* Patients will be instructed to rinse twice daily with a 0.12% chlorhexidine gluconate solution for 2 weeks, and the sutures will be removed after 2 weeks later.
* Analgesic and antibiotic drugs were prescribed after the surgical procedure. Ibobrufen (400 mg.) will be prescribed upon patient's need with a maximum dose 2400mg per day for pain relief [40]. Amoxicillin (500 mg.) every 12 hours for 7 days or clindamycin (300 mg.) every 8 hours for 5 days, for patients having a penicillin allergy, three times per day, for infection control [41].

  5. Assessment:

A) Clinical assessment:

1. Dimensional changes width changes will be measured using bone caliper at baseline immediately following tooth extraction and 4 months postoperatively [42].
2. Postoperative Pain level Pain score will be reported by the patient directly through Visual Analogue Scale score (between 0 and 10. 0: no pain, 1: minimal pain, 5: moderate pain, 10: severe pain) VAS will be recorded at day 14 post-extraction [43]. Post-operative pain was assessed indirectly by mean consumption of analgesics for 7 days postoperatively, will be recorded in milligrams[44].
3. Postoperative wound healing Wound healing will be recorded the 1st and 2 weeks postoperatively through Landry Wound Healing Index (LWHI) [45] which evaluates the extraction site based on tissue color, response to touch, the marginality of the incision line, and extent of the area. The rating is from 1 = very poor to 5 = excellent.

B) Radiographic assessment:

Dimensional changes will be measured using Cone Beam computed Tomography (CBCT) at baseline immediately following tooth extraction and 4 months postoperatively [42].

C) Histomorphometric assessment:

Histological and histomorphometric assessment of bone regeneration patterns of core biopsy harvested at the re-entry surgery for implant placement 4 months post extraction using H&E stains to evaluate bone trabeculae and Modified Masson Trichrome to evaluate bone maturity[46].

ELIGIBILITY:
Inclusion Criteria:

1. Age range (18-40).
2. Hopeless teeth indicated for extraction such as root fractures, caries, internal root resorption, external root resorption, endodontic failures.
3. Systemically free patients using Cornell Medical Index-Health Questionnaire [36].
4. Patients diagnosed with intact surrounding alveolar bone (socket type I) [37].
5. Maxillary anterior teeth and/or premolars indicated for extraction.
6. Enough zone of keratinized tissue (≥2 mm).

Exclusion Criteria:

1. Smokers
2. Occlusal trauma at the site of the graft
3. Pregnancy and lactation
4. Bad compliance with the plaque control instructions following initial therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Dimensional changes | six months
  Clinical measurement using bone caliper. Radiographic measurement using CBCT

SECONDARY OUTCOMES:
Postoperative Pain level Postoperative wound Healing Patterns of bone regeneration of extraction socket | six months
  Visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
depends on publication requirment at publishing status

REFERENCES:
- [Result] Atwood DA. Some clinical factors related to rate of resorption of residual ridges. 1962. J Prosthet Dent. 2001 Aug;86(2):119-25. doi: 10.1067/mpr.2001.117609. No abstract available. PMID 11514795